CLINICAL TRIAL: NCT04099823
Title: MR Evaluation of Cerebrospinal Fluid (CSF) Dynamics and Association of Intracranial CSF Flow With Brain Function
Brief Title: MR Evaluation of Cerebrospinal Fluid (CSF) Dynamics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Petrice M. Cogswell, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-005910
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Hydrocephalus; Alzheimer Disease
MeSH Terms: conditions — Hydrocephalus; Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MR brain (Other): Participants will be asked to complete a MRI screening form to check for the presence of metallic implants and materials. People with pacemakers, aneurysm clips, and cochlear implants, or metal/foreign objects in their eyes cannot have an MRI and will not be able to participate in the study.
  Pre-menopausal females will be asked if they think they may be pregnant. If yes, a urine pregnancy test will be performed.
  Those who meet eligibility criteria for the study and have agreed to participate will be taken to the MRI suite when MR imaging of the brain will be performed.
  Interventions: Other: MRI screening form; Diagnostic Test: Urine pregnancy test; Diagnostic Test: MR brain

INTERVENTIONS:
Other: MRI screening form — Participants will be asked to complete a MRI screening form to check for the presence of metallic implants and materials. People with pacemakers, aneurysm clips, and cochlear implants, or metal/foreign objects in their eyes cannot have an MRI and will not be able to participate in the study.
Diagnostic Test: Urine pregnancy test — Pre-menopausal females will be asked if they think they may be pregnant. If yes, a urine pregnancy test will be performed.
Diagnostic Test: MR brain — You will be asked to lie down on the bed of the MRI scanner. Then a MRI coil/"antenna" will be placed over your head. This will allow us to get clearer pictures of the tissue of interest. The MRI machine makes loud knocking sounds. Because of this you will be asked to wear earplugs. You will receive a "squeeze ball" alarm in case you need urgent help. We will be able to talk with you and hear you during the MRI exam. The entire MRI scan will last about 45-60 minutes. The MR exam will include standard clinical images as well as the CSF flow imaging.

SUMMARY:
The Researchers are trying to test a MR imaging method for detection of Cerebral Spinal Fluid (CSF) flow in the brain to help diagnosis and better understand diseases that affect brain function.

DETAILED DESCRIPTION:
The purpose of this research is to figure out if MR imaging can detect movement of CSF (fluid around the brain) to help better diagnosis and understand the cause of diseases that affect brain function. We are doing this research study to find out if movement of CSF is different between healthy adults and those with a disease that affects brain function.

ELIGIBILITY:
Inclusion Criteria:

* A healthy control will be defined as an otherwise healthy person who does not have a medical condition that affects brain function or have problems with concentration, memory, balance, or coordination.
* Patients who have a suspected diagnosis of altered CSF dynamics including but not limited to normal pressure hydrocephalus will be referred to Dr. Cogswell by their care team to be included in the study. Conditions of altered CSF dynamics include obstructive and non-obstructive hydrocephalus and may be associated with headaches and/or decreased cognitive function.
* Similarly, patients with impaired cognitive function including but not limited to Alzheimer's disease will be referred to Dr. Cogswell by their care team to be included in the study.

Exclusion Criteria:

* Subjects with non-MRI compatible devices
* required sedation
* women who may be pregnant will be excluded.
* The first 10 subjects with normal pressure hydrocephalus will not have previously been shunted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
CSF flow measurement | At the time of MR exam, approximately one hour
  CSF flow will be measured in participants and compared between those with unimpaired brain function and those with clinical diagnosis of a disease that affects brain function, such as Alzheimer's disease and normal pressure hydrocephalus.

SECONDARY OUTCOMES:
Volume of CSF spaces | At the time of MR exam, approximately one hour
  Using standard clinical imaging techniques and computer-automated segmentation methods, the intra and extra-ventricular CSF volume will be measured for each subject.
White matter disease | At the time of MR exam, approximately one hour
  Using standard clinical imaging techniques and computer-automated algorithms, the volume of white matter disease (hyperintense foci in the white matter on T2-weighted MR sequences) will be measured in each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Petrice Cogswell, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials